CLINICAL TRIAL: NCT02645877
Title: Ten-year Trends in the Pre-hospital Emergency Care Spectrum in Beijing From 2005 to 2014: A Multicenter, Retrospective, Observational Study
Brief Title: Trends of the Pre-hospital Emergency Care Spectrum in Beijing From 2005 to 2014: A Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Emergency Medical Center (Other); Beijing Red Cross Emergency Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: PUPH-DTO-201501
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Emergencies [Disease/Finding]
Keywords: Pre-hospital Care; Diseases Spectrum; Call Demands; Emergency Response Time
MeSH Terms: conditions — Emergencies | interventions — Emergency Medical Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prehospital care: All pre-hospital service data were collected from January 2005 to December 2014 from the Beijing Emergency Center and Beijing Red Cross Emergency Center, which oversee all pre-hospital care in Beijing. The major illnesses were classified into 34 disease spectrum categories according to the Medical Priority Dispatch System (MPDS) which total includes 34 diseases. Data on pre-hospital emergency demand and first aid-related time intervals were analyzed to determine trends over the period.
  Interventions: Procedure: Prehospital care

INTERVENTIONS:
Procedure: Prehospital care — The common cause of pre-hospital care demands were Abdominal Problems, Allergies/Envenomation, Animal Bites, Assault/Sexual, Back Pain, Breathing Problems, Burns/Explosions, Carbon Monoxide/Inhalation/Radiation/Hazardous Material, Cardiac or Respiratory Arrest, Chest Pain, Choking, Convulsions/Seizures, Diabetic Problems, Drowning/Diving/Scuba Accident, Electrocution/Lightning, Eye Problems/Injuries, Falls, Headache, Heart Problems, Heat/Cold Exposure, Hemorrhage/Lacerations, Inaccessible Incident/Entrapments, Overdose/Poisoning, Pregnancy/Childbirth/Miscarriage, Psychiatric/Suicide Attempt, Sick Person, Stabbing/Gunshot/Penetrating Trauma, Stroke, Traffic Injuries, Traumatic Injuries, Unconscious/Fainting, Unknown Problems, Inter-Facility Transfer/Palliative Care, Flu-Like Symptoms, etc.

SUMMARY:
This was a retrospective analysis of a cohort of all emergency care patients in Beijing from January 2005 to December 2014. This aim of this study was to analyze the trends in pre-hospital emergency care need and the emergency response times, with the intention of aiding the government to optimize medical resources and improve pre-hospital emergency care.

DETAILED DESCRIPTION:
Pre-hospital emergency care is a very important part of Emergency Medical Service (EMS) System, crucial to patients' life support, disability and mortality rate reduction. The level of pre-hospital emergency care reflects the comprehensive ability of the organizational, management and public welfare of a country. Beijing Emergency Center and Beijing Red Cross Emergency Center are in the charge of all the pre-hospital emergency care in Beijing, which respectively subordinate to Beijing government and Chinese Red Cross Society. This study collected the data of 3,909,746 cases from these two pre-hospital care centers from January, 2005 to December, 2014 and retrospective analyzed the pre-hospital emergency call demand and first aid related time. The results of this study can help the government optimize medical resources; strengthen the prevention of related emergency diseases. The changes and trends of pre-hospital care disease spectrum also present the same problems and situation of developing megacities like Beijing. Based on the meticulous work in these 2 centers, this study has collected the most complete pre-hospital emergency care data in China.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated by pre-hospital care from the Beijing Emergency Medical Center and Beijing Red Cross Emergency Center from January 2005 to December 2014

Exclusion Criteria:

* missing data
* duplicate records
* no identifiable chief cause cases
* not emergency cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pre-hospital service data from the Beijing Emergency Medical Center and Beijing Red Cross Emergency Center were collected from January 2005 to December 2014.
Sampling Method: Non-Probability Sample
Enrollment: 3909746 (Actual)
Dates: Start 2005-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cause of the emergency | 10 years
  The chief complaints of the patients were classified into 34 illnesses according to the Medical Priority Dispatch System (MPDS) which total includes 34 diseases.

SECONDARY OUTCOMES:
The pre-hospital emergency call demand | 10 years
  Total number of pre-hospital emergency calls, reduces the number of missing record, records with no identifiable chief complaint, repeated data, not-emergency care.
Emergency care-related time | 10 years
  Emergency care-related time included emergency response time (ERT), active response time (ART), and passive response time (PRT). ART was defined as the time from emergency call to ambulance departure time; PRT was from departure time to arrival time at the pre-hospital center; ERT was the time from the emergency call to arrival time.

CONTACTS AND LOCATIONS:
Overall Officials: Baoguo Jiang, MD, PhD, Study Chair — Peking University, People's Hospital, Beijing, China
Locations (2):
- China (2):
  - Beijing Emergency Center, Beijing, China, Beijing, Beijing Municipality
  - Beijing Red Cross Emergency center, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang T, Yin X, Zhang P, Kou Y, Jiang B. Road traffic injury and rescue system in China. Lancet. 2015 Apr 25;385(9978):1622. doi: 10.1016/S0140-6736(15)60794-2. No abstract available. PMID 25943819